CLINICAL TRIAL: NCT04329702
Title: Optimizing a Self-directed Mobile Coping Skills Training Intervention to Improve Cardiorespiratory Failure Survivors' Psychological Distress
Brief Title: Mobile Coping Skills Training to Improve Cardiorespiratory Failure Survivors' Psychological Distress
Acronym: Blueprint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00101848; 1R34HL145387 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-12

CONDITIONS: Cardiorespiratory Failure
Keywords: cardiorespiratory failure; critical illness; psychological distress; depression; intensive care units; adults; mechanical ventilation; post-traumatic stress disorder; anxiety
MeSH Terms: conditions — Critical Illness; Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized control clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI and analysts blinded to allocation. Outcomes completed by participants via a mobile app and as such, outcomes assessors are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- coping skills training plus therapist input (Experimental): Participants will receive a CST therapist call within 48 hours of randomization to discuss the study rationale, to conduct a relaxation exercise, and to review app and study logistics. Participants will use the Blueprint mobile app for 1 month.
  Interventions: Behavioral: Coping skills training mobile app with call from CST therapist
- coping skills training without therapist input (Experimental): Participants will receive a call from a research coordinator to get them started with the trial. Participants will use the Blueprint mobile app for 1 month. No therapist calls will be provided. Chat room access in the app will be provided.
  Interventions: Behavioral: Coping skills training mobile app only
- usual care control (No Intervention): Control participants will receive the same safety oversight as intervention participants and will be provided with phone and email contacts for study staff.

INTERVENTIONS:
Behavioral: Coping skills training mobile app with call from CST therapist — The intervention is a mobile app that delivers a 4-week long program of coping skills training. The app contains video, visual, and text content and has a companion PDF workbook. It provides timeline-driven prompts to complete weekly tasks (e.g., viewing videos, completing surveys) and coaching participants to use their current stressors as context for real-life application of adaptive coping skills. A therapist will call participant to introduce the intervention and perform a brief relaxation exercise.
  Other Names: Blueprint; mobile coping skills training (mCST) plus therapist
  Arms: coping skills training plus therapist input
Behavioral: Coping skills training mobile app only — The intervention is a mobile app that delivers a 4-week long program of coping skills training. The app contains video, visual, and text content and has a companion PDF workbook. It provides timeline-driven prompts to complete weekly tasks (e.g., viewing videos, completing surveys) and coaching participants to use their current stressors as context for real-life application of adaptive coping skills. App chat room access will be provided.
  Other Names: Blueprint; mobile coping skills training (mCST)
  Arms: coping skills training without therapist input

SUMMARY:
This is a pilot randomized clinical trial involving adult survivors of cardiorespiratory failure treated in intensive care units (ICUs) that is designed to test the acceptability, feasibility, and clinical impact of a coping skills training intervention (Blueprint) delivered via a mobile app. This trial will allow us to determine if new changes to intervention delivery, inclusion criteria, and other factors are successful. It will also inform the development of a next-step efficacy focused trial.

DETAILED DESCRIPTION:
As survival has improved for the 2 million people with cardiorespiratory failure managed annually in US intensive care units (ICUs), research has clarified how these survivors suffer from severe and persistent symptoms of psychological distress-depression, anxiety, and post-traumatic stress disorder (PTSD)-after discharge. However, few interventions exist that are relevant to patients' experiences and that also accommodate their many physical, social, and financial barriers to personalized care. To fill this gap, we developed a telephone- and web-based coping skills training (CST) program.

CST is an empirically-supported psychosocial intervention that targets the use of the adaptive coping skills to decrease psychological distress and improve quality of life. We conducted a multicenter randomized clinical trial (RCT) called CSTEP that compared CST to an education program (EP) among a general sample of ICU survivors who received mechanical ventilation for cardiorespiratory failure. CST reduced depression symptoms and improved quality of life at 6 months in a pre-specified subgroup with elevated baseline distress. This RCT also identified key questions regarding best practices for identifying patients who are highly distressed yet whose physical illness is manageable, as well as delivering the intervention in a more convenient, and scalable manner. In a recent RCT testing a mindfulness intervention (LIFT), we found that a self-directed mobile app approach increased dose, adherence, and retention. However, many patients reported low enthusiasm for a meditation-based intervention.

What is needed before a second multicenter RCT is to apply the promising CST content to a LIFT-inspired mobile app-based delivery system, and then to test it within a targeted patient population with a high likelihood of response (i.e., high baseline psychological distress). Therefore, we propose a 2-year R34 mixed-methods project that includes a pilot RCT in which we will randomize 45 cardiorespiratory failure / insufficiency survivors to one of three arms in equal ratios: intervention plus therapist for non-responders (n ~15), intervention without a therapist (n ~15), and usual care control (n ~15). Randomization will be stratified by ICU service (medical vs. surgical), baseline HADS score (<14 vs. ≥14), and age (<50 vs. ≥50). Our specific aims will: (1) Optimize the usability of a self-directed mobile app (Blueprint) and an automated post-discharge distress screening system; (2) Test two promising iterations of Blueprint vs. usual care in a pilot 3-arm RCT with 3-month follow up, and (3) Explore facilitators and barriers to Blueprint implementation, using these data to inform any necessary final revisions to the Blueprint app.

ELIGIBILITY:
INCLUSION CRITERIA

1. Adult (age ≥18)
2. Managed in a hospital setting for ≥24 hours during the time inclusion criterion #3 is met.
3. Acute cardiorespiratory failure / insufficiency, defined as ≥1 of the following:

   * mechanical ventilation via endotracheal tube for ≥4 hours
   * non-invasive ventilation (CPAP, BiPAP) for ≥4 hours in a 24-hour period provided for acute respiratory failure
   * new use of supplemental oxygen ≥2 liters per minute (or increase in baseline continuous oxygen)
   * use of vasopressors for shock of any etiology
   * use of inotropes for shock of any etiology
   * use of pulmonary vasodilators
   * use of aortic balloon pump or cardiac assist device for cardiogenic shock
   * use of diuretic intravenous drip
4. Cognitive status intact

   * No history of pre-existing significant cognitive impairment (e.g., dementia) as per medical chart
   * Absence of current significant cognitive impairment (impairment defined as ≥3 errors on the Callahan cognitive status screen)
   * Decisional capacity present
5. Absence of severe and/or persistent mental illness

   * Treatment for severe and/or persistent mental illness (e.g., psychosis, bipolar affective disorder, schizoaffective disorder, schizoid personality disorder, schizophrenia [as per medical record], hospitalization for any psychiatric disorder) within the 6 months preceding the current hospital admission
   * No endorsement of active suicidality at time of admission or informed consent
   * No active substance abuse at a severity that impairs ability to participate
6. Functional English fluency

EXCLUSION CRITERIA (in hospital):

1. Complex medical care expected soon after discharge (e.g., planned surgeries, transplantation evaluation, extensive travel needs for follow up care, disruptive chemotherapy/radiation regimen)
2. Unable to complete study procedures as determined by staff
3. Lack of access to either reliable smartphone with cellular data plan or wifi

INCLUSION CRITERIA (post-discharge)

1. Elevated baseline (T1) psychological distress symptoms, defined as HADS total score of ≥8

EXCLUSION CRITERIA (post-discharge)

1. Failure to randomize within 2 months post-discharge.
2. Failure to access app within 1 month after randomization in the absence of other explanation (e.g., hospitalization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will follow all NIH guidelines and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will follow NIH and institutional guidelines.
Access Criteria: We will follow NIH and institutional guidelines.

REFERENCES:
- [Background] Cox CE, Hough CL, Carson SS, White DB, Kahn JM, Olsen MK, Jones DM, Somers TJ, Kelleher SA, Porter LS. Effects of a Telephone- and Web-based Coping Skills Training Program Compared with an Education Program for Survivors of Critical Illness and Their Family Members. A Randomized Clinical Trial. Am J Respir Crit Care Med. 2018 Jan 1;197(1):66-78. doi: 10.1164/rccm.201704-0720OC. PMID 28872898
- [Background] Cox CE, Porter LS, Hough CL, White DB, Kahn JM, Carson SS, Tulsky JA, Keefe FJ. Development and preliminary evaluation of a telephone-based coping skills training intervention for survivors of acute lung injury and their informal caregivers. Intensive Care Med. 2012 Aug;38(8):1289-97. doi: 10.1007/s00134-012-2567-3. Epub 2012 Apr 18. PMID 22527082
- [Derived] Cox CE, Kelleher SA, Parish A, Olsen MK, Bermejo S, Dempsey K, Jaggers J, Hough CL, Moss M, Porter LS. Feasibility of Mobile App-based Coping Skills Training for Cardiorespiratory Failure Survivors: The Blueprint Pilot Randomized Controlled Trial. Ann Am Thorac Soc. 2023 Jun;20(6):861-871. doi: 10.1513/AnnalsATS.202210-890OC. PMID 36603136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Started | 16 | 14 | 15
Completed | 13 | 8 | 13
Not Completed | 3 | 6 | 2
Not completed — illness | 3 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control | Total
Number analyzed (Participants) | 16 | 14 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.5) | 52.7 (15.0) | 46.5 (14.1) | 49.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 5 | 27
  Male | 5 | 3 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 16 | 12 | 15 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 7 | 0 | 4 | 11
  White | 9 | 11 | 11 | 31
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 15 | 45
Financial distress [Count of Participants; unit: Participants] | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Questionnaire
Description: Depression and anxiety symptoms. Scores range from 0 (better) to 42 (worse)
Time Frame: Between baseline and 1 month post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 11.7 [8.5 to 14.8] | 11.3 [7.7 to 14.8] | 12.1 [8.7 to 15.6]

2. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Questionnaire
Description: Depression and anxiety symptoms. Scores range from 0 (better) to 42 (worse)
Time Frame: Between baseline and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 11.0 [7.2 to 14.8] | 11.4 [6.8 to 16.1] | 13.5 [9.5 to 17.5]

3. Secondary Outcome: Change in Post-Traumatic Stress Symptom Inventory (PTSS)
Description: Post-traumatic stress disorder symptoms. Scores can range from 10 (best) to 70 (worst).
Time Frame: Between baseline and 1 month post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 28.8 [23.7 to 33.9] | 26.4 [20.6 to 32.1] | 30.5 [25.0 to 36.1]

4. Secondary Outcome: Change in Post-Traumatic Stress Symptom Inventory (PTSS)
Description: Post-traumatic stress disorder symptoms. Scores can range from 10 (best) to 70 (worst).
Time Frame: Between baseline and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 28.9 [22.0 to 35.9] | 29.4 [21.0 to 37.8] | 31.3 [24.2 to 38.4]

5. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: A measure of acceptability. Scores can range from 5 (worst) to 35 (best)
Time Frame: 1 month post-randomization
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 29 [27 to 30] | 29.5 [24 to 32.5] | 25 [23 to 30]

6. Secondary Outcome: Intervention Adherence
Description: Measured by how many total tasks of the 33 possible that participants completed within the app during the intervention. Note that a value >33 indicates that participants completed more tasks than required.
Time Frame: 1 month post-randomization
Population: Participants who received intervention.
Measure: Mean (Standard Deviation); unit: tasks
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 14 | 13 | 0
tasks | 36.5 (11.8) | 34.1 (10.9) |

7. Secondary Outcome: Change in Quality of Life Visual Analog Scale
Description: A measure of quality of life. Scores can range from 0 (worst) to 100 (best)
Time Frame: Between baseline and 1 month post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 54.0 [44.6 to 63.4] | 66.7 [56.0 to 77.4] | 61.8 [51.5 to 72.1]

8. Secondary Outcome: Change in Quality of Life Visual Analog Scale
Description: A measure of quality of life. Scores can range from 0 (worst) to 100 (best)
Time Frame: Between baseline and 3 month post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 61.4 [50.6 to 72.3] | 72.5 [58.3 to 86.7] | 67.1 [55.9 to 78.3]

9. Secondary Outcome: Patient Health Questionnaire 10-item Scale (PHQ-10)
Description: An adapted version of the PHQ-15; a measure of physical symptoms. Scores can range from 0 (best) to 30 (worst).
Time Frame: 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 16 | 14 | 15
units on a scale | 11.3 (2.7) | 10.1 (2.7) | 8.3 (2.9)

10. Secondary Outcome: Patient Health Questionnaire 10-item Scale (PHQ-10)
Description: An adapted version of the PHQ-15; a measure of physical symptoms. Scores can range from 0 (best) to 30 (worst).
Time Frame: 3 months post-randomization
Population: Participants with a PHQ-10 score available at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 13 | 8 | 13
units on a scale | 7.9 (2.8) | 6.5 (3.8) | 5.7 (4.0)

11. Secondary Outcome: Distress Associated With Depression and Anxiety Symptom Frequency
Description: A visual analog scale appended to the HADS which allows participants to report how distressing they perceive the depression and anxiety symptoms to be that they reported in the HADS. Scores range from 0 (best) to 100 (worst)
Time Frame: Between baseline and 1 month post-randomization
Population: Data not collected.
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Distress Associated With Depression and Anxiety Symptom Frequency
Description: as for outcome 11
Time Frame: Between baseline and 3 months post-randomization
Population: Data not collected.
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Distress Associated With PTSD Symptom Frequency
Description: A visual analog scale appended to the PTSS which allows participants to report how distressing they perceive the depression and anxiety symptoms to be that they reported in the PTSS. Scores range from 0 (best) to 100 (worst)
Time Frame: Between baseline and 1 month post-randomization
Population: Data not collected.
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Distress Associated With PTSD Symptom Frequency
Description: as for outcome 13
Time Frame: Between baseline and 3 months post-randomization
Population: Data not collected.
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Coping Skills Training Plus Therapist Input | Coping Skills Training Without Therapist Input | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 2/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04329702/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04329702/SAP_002.pdf
  • Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT04329702/ICF_000.pdf